CLINICAL TRIAL: NCT06735807
Title: Comparing Generated AI (Emohaa) and Group ACT in Reducing Emotional Distress: a Randomized Controlled Trial
Brief Title: Generated AI-informed Intervention (Emohaa) vs Group ACT vs WL on Emotional Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central University of Finance and Economics, China (Other)
Responsible Party: Principal Investigator, Yi Feng, Associate Private Investigator, Central University of Finance and Economics, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CUFE-20240229-0001
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-09

CONDITIONS: Artificial Intelligence (AI); Depression - Major Depressive Disorder; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Generated AI (Emohaa) (Experimental)
  Interventions: Behavioral: Generated AI-based intervention (Emohaa)
- Group ACT (Active Comparator)
  Interventions: Behavioral: group ACT
- Waitlist Group (WLG) (Sham Comparator)
  Interventions: Behavioral: wailist (delayed intervenion)

INTERVENTIONS:
Behavioral: Generated AI-based intervention (Emohaa) — Participants will complete the intervention process by interacting with the Wechat applet. Participants will be required to complete a 6-week self-help therapy. Participants will be required to have a 30-minute dialogue including input and reflection time with Emohaa each week simultaneously with group ACT. Participants are free to dialogue with Emohaa for the rest of the week. An independent research assistant will monitor the intervention process from the platform. If the corresponding dialogue is not completed on time each week, the participant will be reminded via WeChat to complete this session before the start of the next session in the following week.
  Arms: Generated AI (Emohaa)
Behavioral: group ACT — A 6-week group ACT intervention. Each group has 6-10 participants. Each session is one hour.
  Arms: Group ACT
Behavioral: wailist (delayed intervenion) — During the intervention period, participants in the WLG were only required to complete the appropriate assessments without receiving any intervention. Upon completion of the 15-day follow-up assessment, participants in the WLG could be free to choose to receive one of the two interventions. The intervention will be the same as the corresponding experimental group.
  Arms: Waitlist Group (WLG)

SUMMARY:
Emotional Distress, such as anxiety and depression, is an essential issue worldwide. There have been several evidence-based psychotherapies that are effective in improving emotional distress, such as Acceptance and Commitment Therapy (ACT). However, the scarcity of professionals and the imbalance in the distribution of mental health resources prevent individuals in need from accessing immediate and effective help.

Artificial intelligence (AI) has the potential to promote this problem. The existing studies have provided preliminary support for the application of AI in mental health interventions. One such model, Emohaa, a generated AI model, has been examined for its effectiveness in adult emotional distress. However, despite the limited reliability of the single-group design, parallel randomized controlled trials are scarce to validate this finding further. This present study is to fill this gap.

This study aims to examine the effectiveness of the generated AI (Emohaa) in reducing emotional distress, including anxiety and depression, compared with group ACT and waitlist. In this parallel randomized controlled trial, it is hypothesized that (1) Compared with the waitlist, Emohaa and group ACT could significantly improve participants' emotional distress, including anxiety and depression symptoms; (2) Emohaa would lead to a greater reduction in anxiety and depression symptoms compared with group ACT.

ELIGIBILITY:
Inclusion Criteria:

* Adults with 18-25 ages;
* Suffering from emotional distress (PHQ-9 > 9 or GAD-7 > 9);
* Ability to use the mobile phone to interact with AI;
* Consent to participate in the study.

Exclusion Criteria:

* High risk of self-injury and suicide;
* Presence of psychotic symptoms (i.e., delusions);
* Serious substance use problems;
* Other mental or physical illnesses requiring urgent medical assistance;
* Received other psychological or pharmacological interventions in the last month

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 0, 2, 4, 6, 8, and 10 weeks
  PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Generalized Anxiety Disorder (GAD-7) | 0, 2, 4, 6, 8, and 10 weeks
  GAD-7 is an easy-to-perform initial screening tool for generalized anxiety disorder. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
UCLA Loneliness Scale (ULS-3) | 0, 2, 4, 6, 8, and 10 weeks
  ULS-3 is a brief version of the UCLA Loneliness Scale with 3 items, which was designed to assess loneliness. Questions are scored on a Likert scale of 1-4 with 1 being never and 4 being always.
Self-Concept Clarity Scale (SCCS) | 0, 2, 4, 6, 8, and 10 weeks
  SCCS is a 12-item scale to measure the clarity of self-concept. Questions are scored on a Likert scale of 1-5 with 1 being strongly disagree and 5 being strongly agree.
Acceptance and Action Questionnaire-2nd Edition (AAQ-II) | 0, 2, 4, 6, 8, and 10 weeks
  AAQ-II is the second version of the Acceptance and Action Questionnaire with 7 items. Questions are scored on a Likert scale of 1-7 with 1 being never and 7 being always
Insomnia Severity Index (ISI) | 0, 2, 4, 6, 8, and 10 weeks
  ISI is a 7-item screening tool to measure the severity of sleep problems. Questions are scored on a 0-4 scale with different descriptions
Client Satisfaction Questionnaire (CSQ-8) | 2, 4, 6, 8, and 10 weeks
  CSQ-8 is an easy-to-perform initial screening tool for client satisfaction with mental health services. Questions are scored on a Likert scale of 1-4 with 1 being low satisfaction and 4 being high satisfaction.
Digital Working Alliance Inventory (DWAI) | 6, 8, and 10 weeks
  DWAI is an 8-item scale to measure the working alliance between participants and the AI model revised by the Working Alliance Inventory. Questions are scored on a Likert scale of 1-7 with 1 being totally disagree and 7 being totally agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Central University of Finance and Economics, China, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Personal contact in reliable reason
Supporting Information: Analytic Code